CLINICAL TRIAL: NCT00545129
Title: PHASE II RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED MULTICENTER EFFICACY AND SAFETY STUDY OF TANEZUMAB AS ADD-ON THERAPY TO OPIOID MEDICATION IN PATIENTS WITH PAIN DUE TO BONE METASTASES
Brief Title: A Study Of Tanezumab as Add-On Therapy to Opioid Medication In Patients With Pain Due To Cancer That Has Spread To Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091003; 2008-005181-31 (EudraCT Number); CANCER PAIN POC (Other: Alias Study Number)
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Neoplasm Metastasis; Palliative Care
MeSH Terms: conditions — Neoplasm Metastasis | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tanezumab 10 mg IV + opioids (Experimental)
  Interventions: Drug: Tanezumab 10 mg IV
- Placebo + opioids (Placebo Comparator): Single IV infusion of placebo for tanezumab on Day 1. Maintained on baseline opioid regimen.
  Interventions: Drug: IV Placebo for tanezumab

INTERVENTIONS:
Drug: Tanezumab 10 mg IV — Single IV infusion of 10 mg tanezumab on Day 1. Maintained on baseline opioid regimen.
  Arms: Tanezumab 10 mg IV + opioids
Drug: IV Placebo for tanezumab — Single IV infusion of placebo for tanezumab on Day 1. Maintained on baseline opioid regimen.
  Arms: Placebo + opioids

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of tanezumab in combination with opioids in treating pain due to cancer that has spread to bone.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer, breast cancer, renal cell carcinoma or multiple myeloma that has spread to bone, causing moderate to severe bone pain.
* Requires daily opioid medication

Exclusion Criteria:

* Patients who do not have bone pain caused by cancer are not eligible for the study.
* Patients who started chemotherapy less than 4 weeks ago, or who completed radiotherapy less than 4 weeks ago, are not eligible.
* Known history or evidence of osteoarthritis. History of significant trauma to a major joint within 1 year prior to Screening.
* Known history of rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-04-29 (Actual); Primary Completion 2011-12-24 (Actual); Study Completion 2012-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (12):
  - UCSD Center for Pain Medicine, La Jolla, California
  - UCSD Medical Center - Thornton Hospital, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Indiana Pain and Spine Clinic, South Bend, Indiana
  - WK River Cities Clinical Research Center, Shreveport, Louisiana
  - Willis Knighton Pierremont Health Center, Shreveport, Louisiana
  - Hollings Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina, Department of Urology, Charleston, South Carolina
  - MUSC Department of Radiology, Charleston, South Carolina
  - MUSC Investigational Pharmacy, Charleston, South Carolina
  - MUSC Urology Ambulatory Care, Charleston, South Carolina
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
- Austria (3):
  - Landeskrankenhaus Graz - Universitaetsklinik fuer Orthopaedie und Orthopaedische Chirurgie, Graz
  - Krankenhaus der Elisabethinen Linz, Institut fuer Anaesthesiologie und Intensivmedizin, Linz
  - Nuhr Zentrum, Senftenberg
- Bosnia and Herzegovina (2):
  - Clinic of Oncology, Banja Luka
  - Institute of Oncology, University Clinical Center Sarajevo, Sarajevo
- General Hospital Varazdin, Varaždin, Croatia
- Institut Gustave Roussy, Villejuif, France
- Hungary (3):
  - Fovarosi Onkormanyzat Peterfy Sandor Utcai Korhaz - Fajdalom Ambulancia, Budapest
  - Fovarosi Onkormanyzat Jahn Ferenc Del-pesti Korhaz - Fajdalom Ambulancia, Budapest
  - Fejer Megyei Szt. Gyorgy Korhaz - Rendelointezet/Aneszteziologiai es Intenziv Betegellato Osztaly, Székesfehérvár
- India (5):
  - Shri Siddhivinayak Ganpati Cancer Hospital, Miraj, Maharashtra
  - Central India Cancer Research Institute, Nagpur, Maharashtra
  - Shatabdi Superspeciality Hospital, Nashik, Maharashtra
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow, Uttar Pradesh
  - Rajiv Gandhi Cancer Institute and Research Centre,, New Delhi
- 10th Department, Latvian Oncological Centre / Riga Eastern Clinical University Hospital, Riga, Latvia
- Centro de Cancer del Centro Medico ABC, Mexico City, Mexico City, Mexico
- Peru (2):
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima, LIMA L13
  - Oncocare, Lima
- Poland (4):
  - Niepubliczny Zaklad Opieki Zdrowotnej, Bydgoszcz
  - Hospicjum im. Ks. Eugeniusza Dutkiewicza SAC w Gdansku, Gdansk
  - Poradnia Medycyny Paliatywnej, Hospicjum Palium, Poznan
  - NZOZ Zespol Opieki Domowej, Włocławek
- Slovakia (2):
  - Fakultna Nemocnica s Poliklinikou F.D.Roosevelta, Banská Bystrica
  - Narodny onkologicky ustav, Bratislava
- South Korea (2):
  - Severance Hospital, Yonsei University College of Medicine, Yonsei Cancer Center, Seoul
  - Samsung Medical Center, Division of Hematology-Oncology, Department of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sopata M, Katz N, Carey W, Smith MD, Keller D, Verburg KM, West CR, Wolfram G, Brown MT. Efficacy and safety of tanezumab in the treatment of pain from bone metastases. Pain. 2015 Sep;156(9):1703-1713. doi: 10.1097/j.pain.0000000000000211. PMID 25919474
- [Derived] Bapat AA, Hostetter G, Von Hoff DD, Han H. Perineural invasion and associated pain in pancreatic cancer. Nat Rev Cancer. 2011 Sep 23;11(10):695-707. doi: 10.1038/nrc3131. PMID 21941281
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091003&StudyName=A%20Study%20Of%20Tanezumab%20as%20Add-On%20Therapy%20to%20Opioid%20Medication%20In%20Patients%20With%20Pain%20Due%20To%20Cancer%20That%20Has%20Spread%20To%20Bone

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Post Week 8 visit, participants were eligible to rollover to extension study A4091029 (NCT00830180).
Groups:
- Tanezumab: Single intravenous infusion of tanezumab 10 mg over 5 minutes on Day 1, along with background opioid medication administered daily for 113 days. Total daily dose of opioid medication was determined as per accepted clinical guidelines in the opioid adjustment period during pre-treatment phase.
- Placebo: Single intravenous infusion of placebo matched to tanezumab over 5 minutes on Day 1, along with background opioid medication administered daily for 113 days. Total daily dose of opioid medication was determined as per accepted clinical guidelines in the opioid adjustment period during pre-treatment phase.
Period: Overall Study
Arm/Group | Tanezumab | Placebo
Started | 29 | 30
Completed | 12 | 6
Not Completed | 17 | 24
Not completed — Lack of Efficacy | 2 | 5
Not completed — Death | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Rollover to Study A4091029 (NCT00830180) | 9 | 14
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 years | 0 | 0 | 0
  18 to 44 years | 1 | 6 | 7
  45 to 64 years | 15 | 15 | 30
  Greater than or equal to (>=) 65 years | 13 | 9 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Pain Intensity Numeric Rating Scale (NRS) Score at Week 6
Description: Daily average pain was assessed on an 11-point NRS over the past 24 hours (before each specified visit), where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". Lower the score, lesser the pain intensity.
Time Frame: Baseline, Week 6
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Missing values were imputed using baseline observation carried forward (BOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale
  Baseline | 5.4 (1.02) | 5.3 (0.98)
  Change at Week 6 | -1.3 (1.81) | -0.9 (1.52)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Analysis of covariance (ANCOVA) model included treatment and cancer type as fixed effects, baseline value as covariate and study site as random effect. Least squares (LS) mean difference, and corresponding 95% confidence interval (CI) were estimated from ANCOVA model; Test type: Superiority or Other; p = 0.569, ANCOVA; Least Squares (LS) Mean Difference = -0.26, 95% CI 2-sided [-1.18 to 0.66], Standard Error of Mean 0.45

2. Secondary Outcome: Change From Baseline in Daily Average Pain Intensity Numeric Rating Scale (NRS) Score at Weeks 1, 2, 4, 8, 12 and 16
Description: Daily average pain was assessed on an 11-point NRS over the past 24 hours (before each specified visit), where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". Lower the score, lesser pain intensity.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Missing values were imputed using BOCF method. For time points after Week 8, inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale
  Change at Week 1 | -0.8 (0.85) | -0.6 (0.86)
  Change at Week 2 | -0.9 (1.08) | -0.8 (1.33)
  Change at Week 4 | -1.3 (1.58) | -1.2 (1.46)
  Change at Week 8 | -1.4 (1.73) | -0.9 (1.47)
  Change at Week 12 | -1.0 (1.56) | -0.4 (1.29)
  Change at Week 16 | -0.8 (1.47) | -0.4 (1.17)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 1: ANCOVA model included treatment and cancer type as fixed effects, baseline value as covariate and study site as random effect. LS mean difference and corresponding 95% CI were estimated from ANCOVA model; Test type: Superiority or Other; p = 0.581, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.60 to 0.34], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Change at Week 2: ANCOVA model included treatment and cancer type as fixed effects, baseline value as covariate and study site as random effect. LS mean difference and corresponding 95% CI were estimated from ANCOVA model; Test type: Superiority or Other; p = 0.795, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.56 to 0.73], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Change at Week 4: ANCOVA model included treatment and cancer type as fixed effects, baseline value as covariate and study site as random effect. LS mean difference and corresponding 95% CI were estimated from ANCOVA model; Test type: Superiority or Other; p = 0.843, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.76 to 0.93], Standard Error of Mean 0.41
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 8: ANCOVA model included treatment and cancer type as fixed effects, baseline value as covariate and study site as random effect. LS mean difference and corresponding 95% CI were estimated from ANCOVA model; Test type: Superiority or Other; p = 0.292, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-1.34 to 0.42], Standard Error of Mean 0.43

3. Secondary Outcome: Change From Baseline in Daily Worst Pain Intensity Numeric Rating Scale (NRS) Score at Week 1, 2, 4, 6, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: The worst pain was assessed an 11-point NRS over the past 24 hours where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". Lower the score, lesser pain intensity.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Missing values were imputed using BOCF method. For time points after Week 8 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale
  Baseline | 6.3 (1.30) | 6.4 (1.06)
  Change at Week 1 | -0.8 (0.87) | -0.6 (0.85)
  Change at Week 2 | -0.8 (1.32) | -1.0 (1.17)
  Change at Week 4 | -1.2 (1.70) | -1.2 (1.40)
  Change at Week 6 | -1.0 (1.82) | -0.9 (1.52)
  Change at Week 8 | -1.1 (1.77) | -0.9 (1.53)
  Change at Week 12 | -0.7 (1.40) | -0.4 (1.42)
  Change at Week 16 | -0.5 (1.27) | -0.4 (1.16)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.299, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.72 to 0.23], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.519, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.47 to 0.91], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.776, ANCOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-0.74 to 0.98], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 6: ANCOVA model included treatment and cancer type as fixed effects, baseline value as covariate and study site as random effect. LS mean difference and corresponding 95% CI were estimated from ANCOVA model; Test type: Superiority or Other; p = 0.978, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.93 to 0.91], Standard Error of Mean 0.45
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.689, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-1.10 to 0.73], Standard Error of Mean 0.45

4. Secondary Outcome: Change From Baseline in Daily Worst Pain Intensity Numeric Rating Scale (NRS) Score at Week 1, 2, 4, 6, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: The worst pain was assessed on 11-point NRS over the past 24 hours where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The lower the value the lesser pain intensity.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Missing values were imputed using LOCF method. For time points after Week 8 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale
  Baseline | 6.3 (1.30) | 6.4 (1.06)
  Change at Week 1 | -0.8 (0.87) | -0.6 (0.85)
  Change at Week 2 | -0.8 (1.32) | -1.0 (1.17)
  Change at Week 4 | -1.1 (1.80) | -1.3 (1.45)
  Change at Week 6 | -1.0 (1.91) | -1.1 (1.59)
  Change at Week 8 | -1.1 (1.86) | -1.1 (1.68)
  Change at Week 12 | -0.8 (1.86) | -1.3 (2.01)
  Change at Week 16 | -0.7 (1.83) | -1.2 (2.01)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.299, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.72 to 0.23], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.519, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.47 to 0.91], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.618, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.68 to 1.13], Standard Error of Mean 0.44
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.818, ANCOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.85 to 1.07], Standard Error of Mean 0.47
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.819, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS Mean Difference = 0.11, 95% CI 2-sided [-0.87 to 1.09], Standard Error of Mean 0.48

5. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Average Pain Scores at Week 1, 2, 4, 6, 8, 12 and 16: BOCF
Description: BPI-sf: self-administered questionnaire developed to assess severity, impact of pain on daily functions, consisted of 5 questions. Questions 1-4 measured magnitude of pain at its worst, least, average, right now. BPI-sf average pain measured the severity of pain based on the average pain experienced over the past 24-hours and ranged from 0 (No Pain) to10 (Pain as bad as you can imagine), lower scores indicates lesser pain intensity. Question 5: 7 item subsets that measured level of interference of pain on daily functions on 11-point NRS at 0 (Does not interfere) to 10 (Completely interferes).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Here "overall number of participants analyzed signifies those participants who were evaluable for this measure. For time points after Week 8 inferential statistics were not performed because post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 27
unit on a scale
  Baseline | 5.2 (1.15) | 5.1 (1.14)
  Change at Week 1 | -0.4 (1.65) | -0.4 (1.12)
  Change at Week 2 | -0.9 (1.99) | -0.8 (1.15)
  Change at Week 4 | -1.0 (1.97) | -1.0 (1.84)
  Change at Week 6 | -1.0 (1.54) | -0.9 (1.78)
  Change at Week 8 | -1.0 (1.43) | -0.9 (1.84)
  Change at Week 12 | -0.9 (1.17) | -0.5 (1.40)
  Change at Week 16 | -0.7 (1.39) | -0.4 (1.22)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.906, ANCOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.66 to 0.74], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.906, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.95 to 0.85], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.613, ANCOVA; LS Mean Difference = 0.26, 95% CI 2-sided [-0.78 to 1.29], Standard Error of Mean 0.50
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.988, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.95 to 0.94], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.922, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-1.01 to 0.92], Standard Error of Mean 0.47

6. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Average Pain Scores at Week 1, 2, 4, 6, 8, 12 and 16: LOCF
Description: BPI-sf: self-administered questionnaire developed to assess severity, impact of pain on daily functions, consisted of 5 questions. Questions 1-4 measured magnitude of pain at its worst, least, average, right now. BPI-sf average pain measured the severity of pain based on the average pain experienced over the past 24-hours and ranged from 0 (No Pain) to 10 (Pain as bad as you can imagine), lower score indicates lesser pain intensity. Question 5: 7 item subsets that measured level of interference of pain on daily functions on 11-point numeric rating scale at 0 (Does not interfere) to 10 (Completely interferes).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Here, overall number of participants analyzed=participants who were evaluable for this measure. number analyzed=participants evaluable at specific time points. For time points after Week 8 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 27
unit on a scale
  Baseline | 5.2 (1.15) | 5.1 (1.14)
  Change at Week 1: number analyzed (Participants) | 20 | 21
  Change at Week 1 | -0.6 (1.90) | -0.5 (1.25)
  Change at Week 2: number analyzed (Participants) | 24 | 25
  Change at Week 2 | -1.0 (2.12) | -1.0 (1.32)
  Change at Week 4: number analyzed (Participants) | 25 | 26
  Change at Week 4 | -1.0 (2.03) | -1.0 (1.87)
  Change at Week 6: number analyzed (Participants) | 25 | 26
  Change at Week 6 | -0.9 (2.00) | -1.1 (1.83)
  Change at Week 8: number analyzed (Participants) | 25 | 26
  Change at Week 8 | -1.6 (1.44) | -1.0 (1.89)
  Change at Week 12: number analyzed (Participants) | 25 | 26
  Change at Week 12 | -1.4 (1.29) | -1.0 (1.95)
  Change at Week 16: number analyzed (Participants) | 25 | 26
  Change at Week 16 | -1.4 (1.55) | -1.0 (1.92)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.655, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-1.03 to 0.66], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.897, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.85 to 0.96], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.798, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.93 to 1.20], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.672, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.83 to 1.27], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.243, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-1.56 to 0.41], Standard Error of Mean 0.48

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Worst Pain Scores at Week 1, 2, 4, 6, 8, 12 and 16: BOCF
Description: BPI-sf: self-administered questionnaire developed to assess severity, impact of pain on daily functions, consisted of 5 questions. Questions 1-4 measured magnitude of pain at its worst, least, average, right now. BPI-sf worst pain measured the severity of pain based on the worst pain experienced over the past 24-hours and ranged from 0 (No Pain) to 10 (Pain as bad as you can imagine), lower scores =lesser pain intensity. Question 5: 7 item subsets that measured level of interference of pain on daily functions on 11-point numeric rating scale at 0 (Does not interfere) to 10 (Completely interferes).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Missing values were imputed using BOCF method. Here overall number of participants analyzed signifies those participants who were evaluable for this measure. For time points after Week 8 inferential statistics were not performed because post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 27
units on a scale
  Baseline | 6.1 (1.54) | 6.0 (1.09)
  Change at Week 1 | -0.8 (1.76) | -0.4 (1.42)
  Change at Week 2 | -1.0 (1.74) | -1.0 (1.74)
  Change at Week 4 | -1.2 (2.01) | -0.8 (1.92)
  Change at Week 6 | -0.7 (2.02) | -0.7 (2.25)
  Change at Week 8 | -1.1 (2.09) | -0.7 (1.98)
  Change at Week 12 | -0.4 (1.48) | -0.7 (1.77)
  Change at Week 16 | -0.5 (1.09) | -0.6 (1.34)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.445, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-1.16 to 0.52], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.992, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-1.00 to 1.00], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.655, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-1.34 to 0.86], Standard Error of Mean 0.53
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.860, ANCOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-1.09 to 1.30], Standard Error of Mean 0.58
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.595, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-1.52 to 0.89], Standard Error of Mean 0.59

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Worst Pain Scores Weeks 1, 2, 4, 6, 8, 12 and 16: LOCF
Description: BPI-sf: self-administered questionnaire developed to assess severity, impact of pain on daily functions, consisted of 5 questions. Questions 1-4 measured magnitude of pain at its worst, least, average, right now. BPI-sf worst pain measured the severity of pain based on the worst pain experienced over the past 24-hours and ranged from 0 (No Pain) to 10 (Pain as bad as you can imagine), lower scores=lesser pain intensity. Question 5: 7 item subsets that measured level of interference of pain on daily functions on11-point numeric rating scale at 0 (Does not interfere) to 10 (Completely interferes).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Overall number of participants analyzed=participants who were evaluable for this measure; number analyzed=participants evaluable at specific time points. For time points after Week 8 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 27
units on a scale
  Baseline | 6.1 (1.54) | 6.0 (1.09)
  Change at Week 1: number analyzed (Participants) | 20 | 21
  Change at Week 1 | -1.1 (1.99) | -0.5 (1.60)
  Change at Week 2: number analyzed (Participants) | 24 | 25
  Change at Week 2 | -1.1 (1.82) | -1.3 (1.86)
  Change at Week 4: number analyzed (Participants) | 25 | 26
  Change at Week 4 | -1.3 (2.06) | -0.9 (1.95)
  Change at Week 6: number analyzed (Participants) | 25 | 26
  Change at Week 6 | -1.1 (2.42) | -1.0 (2.32)
  Change at Week 8: number analyzed (Participants) | 25 | 26
  Change at Week 8 | -1.6 (2.33) | -1.0 (2.11)
  Change at Week 12: number analyzed (Participants) | 25 | 26
  Change at Week 12 | -1.2 (2.33) | -1.1 (2.44)
  Change at Week 16: number analyzed (Participants) | 25 | 26
  Change at Week 16 | -1.2 (2.33) | -1.0 (2.32)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.179, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-1.76 to 0.35], Standard Error of Mean 0.50
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.938, ANCOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-1.02 to 1.10], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.621, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-1.41 to 0.86], Standard Error of Mean 0.55
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.863, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-1.44 to 1.21], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.237, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.95 to 0.51], Standard Error of Mean 0.59

9. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 30 Percent (%), >=50%, >=70% and >=90% Reduction in Daily Average Pain Intensity Numeric Rating Scale (NRS) Score: BOCF
Description: Percentage of participant with response as defined by a >=30%, >=50%, >=70%, and >=90%, reduction in the daily average pain intensity NRS score from baseline, that was maintained for a minimum of 3 consecutive days following this original study day (reduction in pain was maintained for a minimum duration of 4 consecutive days). Daily average pain was assessed on 11-point NRS over the past 24 hours where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". Lower scores indicate less pain intensity.
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Missing values were imputed using BOCF method. Data was not summarized statistically at week 12 and 16 because post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
percentage of participants
  Week 1: >=30% reduction | 10.3 | 13.3
  Week 1: >=50% reduction | 3.4 | 0.0
  Week 1: >=70% reduction | 0.0 | 0.0
  Week 1: >=90% reduction | 0.0 | 0.0
  Week 2: >=30% reduction | 24.1 | 26.7
  Week 2: >=50% reduction | 6.9 | 10.0
  Week 2: >=70% reduction | 0.0 | 0.0
  Week 2: >=90% reduction | 0.0 | 0.0
  Week 4: >=30% reduction | 44.8 | 36.7
  Week 4: >=50% reduction | 27.6 | 16.7
  Week 4: >=70% reduction | 3.4 | 6.7
  Week 4: >=90% reduction | 0.0 | 0.0
  Week 6: >=30% reduction | 14.4 | 33.3
  Week 6: >=50% reduction | 27.6 | 20.0
  Week 6: >=70% reduction | 6.9 | 3.3
  Week 6: >=90% reduction | 0.0 | 3.3
  Week 8: >=30% reduction | 48.3 | 20.0
  Week 8: >=50% reduction | 34.5 | 16.7
  Week 8: >=70% reduction | 6.9 | 6.7
  Week 8: >=90% reduction | 0.0 | 6.7
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 1 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.10 to 4.94]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 2 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.23 to 3.32]
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 2 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.05 to 6.35]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 4 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.601, Fisher Exact; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.44 to 4.53]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 4 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.360, Fisher Exact; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.46 to 8.51]
Statistical Analysis 6: Comparison: Tanezumab vs Placebo; Week 4 (>=70%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.01 to 10.24]
Statistical Analysis 7: Comparison: Tanezumab vs Placebo; Week 6 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.596, Fisher Exact; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.43 to 4.66]
Statistical Analysis 8: Comparison: Tanezumab vs Placebo; Week 6 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.552, Fisher Exact; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.39 to 6.24]
Statistical Analysis 9: Comparison: Tanezumab vs Placebo; Week 6 (>=70%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.612, Fisher Exact; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.10 to 131.03]
Statistical Analysis 10: Comparison: Tanezumab vs Placebo; Week 6 (>=90%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 19.66]
Statistical Analysis 11: Comparison: Tanezumab vs Placebo; Week 8 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.029, Fisher Exact; Odds Ratio (OR) = 3.73, 95% CI 2-sided [1.04 to 14.32]
Statistical Analysis 12: Comparison: Tanezumab vs Placebo; Week 8 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.143, Fisher Exact; Odds Ratio (OR) = 2.63, 95% CI 2-sided [0.67 to 11.36]
Statistical Analysis 13: Comparison: Tanezumab vs Placebo; Week 8 (>=70%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.07 to 15.25]
Statistical Analysis 14: Comparison: Tanezumab vs Placebo; Week 8 (>=90%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.492, Fisher Exact; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 3.57]

10. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 30 Percent (%), >=50%, >=70% and >=90% Reduction in Daily Average Pain Intensity Numeric Rating Scale (NRS) Score: LOCF
Description: as for outcome 9
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Missing values were imputed using LOCF method. Data was not summarized statistically at week 12 and 16 because post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
percentage of participants
  Week 1: >=30% reduction | 10.3 | 13.3
  Week 1: >=50% reduction | 3.4 | 0.0
  Week 1: >=70% reduction | 0.0 | 0.0
  Week 1: >=90% reduction | 0.0 | 0.0
  Week 2: >=30% reduction | 24.1 | 26.7
  Week 2: >=50% reduction | 6.9 | 10.0
  Week 2: >=70% reduction | 0.0 | 0.0
  Week 2: >=90% reduction | 0.0 | 0.0
  Week 4: >=30% reduction | 44.8 | 40.0
  Week 4: >=50% reduction | 27.6 | 16.7
  Week 4: >=70% reduction | 3.4 | 6.7
  Week 4: >=90% reduction | 0.0 | 0.0
  Week 6: >=30% reduction | 41.4 | 40.0
  Week 6: >=50% reduction | 27.6 | 23.3
  Week 6: >=70% reduction | 6.9 | 3.3
  Week 6: >=90% reduction | 0.0 | 3.3
  Week 8: >=30% reduction | 48.3 | 30.0
  Week 8: >=50% reduction | 34.5 | 23.3
  Week 8: >=70% reduction | 6.9 | 6.7
  Week 8: >=90% reduction | 0.0 | 6.7
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 1 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.10 to 4.94]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 2 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.23 to 3.32]
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 2 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.05 to 6.35]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 4 (>=30%) reduction: odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.795, Fisher Exact; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.38 to 3.88]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 4 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.360, Fisher Exact; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.46 to 8.51]
Statistical Analysis 6: Comparison: Tanezumab vs Placebo; Week 4 (>=70%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.01 to 10.24]
Statistical Analysis 7: Comparison: Tanezumab vs Placebo; Week 6 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.33 to 3.39]
Statistical Analysis 8: Comparison: Tanezumab vs Placebo; Week 6 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.771, Fisher Exact; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.33 to 4.83]
Statistical Analysis 9: Comparison: Tanezumab vs Placebo; Week 6 (>=70%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.612, Fisher Exact; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.10 to 131.03]
Statistical Analysis 10: Comparison: Tanezumab vs Placebo; Week 6 (>=90%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 19.66]
Statistical Analysis 11: Comparison: Tanezumab vs Placebo; Week 8 (>=30%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.187, Fisher Exact; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.66 to 7.30]
Statistical Analysis 12: Comparison: Tanezumab vs Placebo; Week 8 (>=50%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.399, Fisher Exact; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.48 to 6.43]
Statistical Analysis 13: Comparison: Tanezumab vs Placebo; Week 8 (>=70%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 1.000, Fisher Exact; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.07 to 15.25]
Statistical Analysis 14: Comparison: Tanezumab vs Placebo; Week 8 (>=90%) reduction: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.492, Fisher Exact; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 3.57]

11. Secondary Outcome: Average Daily Opioid Consumption
Description: The average daily opioid consumption was calculated as the daily sum of total opioid dosage in milligrams. Opioid consumption on each day was converted to the morphine equivalent dosage (MED). Results were summarized for opioid dose adjust period, baseline assessment period and post-baseline period.
Time Frame: Opioid Dose Adjust Period (Day-30 to Day-4), Baseline Assessment period (Day-3 to Day-1), Post Baseline Period (Day 1 to Week 16)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). 'number analyzed'=participants evaluable at specific time period.
Measure: Mean (Standard Deviation); unit: MED
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
MED
  Opioid Dose Adjust Period: number analyzed (Participants) | 28 | 27
  Opioid Dose Adjust Period | 112.8 (123.22) | 98.3 (107.42)
  Baseline Assessment Period | 111.8 (134.59) | 102.0 (112.78)
  Post Baseline Period | 111.9 (137.22) | 102.7 (111.83)

12. Secondary Outcome: Number of Doses of Rescue Medication Required Per Week
Description: Participants received immediate release (IR) opioid as rescue medication as needed for breakthrough pain from Day 1-113 at the dose determined during the pre-treatment phase, provided the average total daily dose of opioids between study visits does not exceed the baseline total daily opioid dose by more than 10%.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: doses per week
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 26 | 21
doses per week
  Week 1 | 9.5 (16.16) | 5.6 (6.21)
  Week 2: number analyzed (Participants) | 25 | 20
  Week 2 | 9.0 (16.57) | 5.0 (6.24)
  Week 3: number analyzed (Participants) | 25 | 19
  Week 3 | 8.9 (17.46) | 5.2 (6.88)
  Week 4: number analyzed (Participants) | 24 | 20
  Week 4 | 9.0 (17.24) | 6.6 (10.82)
  Week 5: number analyzed (Participants) | 23 | 20
  Week 5 | 5.5 (5.62) | 7.1 (10.47)
  Week 6: number analyzed (Participants) | 22 | 20
  Week 6 | 4.8 (5.59) | 8.0 (11.25)
  Week 7: number analyzed (Participants) | 22 | 18
  Week 7 | 5.9 (5.96) | 9.0 (12.49)
  Week 8: number analyzed (Participants) | 22 | 18
  Week 8 | 5.8 (6.08) | 9.9 (12.04)
  Week 9: number analyzed (Participants) | 18 | 15
  Week 9 | 5.2 (5.61) | 3.8 (4.23)
  Week 10: number analyzed (Participants) | 17 | 6
  Week 10 | 11.0 (23.22) | 3.3 (3.98)
  Week 11: number analyzed (Participants) | 16 | 6
  Week 11 | 12.1 (23.75) | 4.7 (5.50)
  Week 12: number analyzed (Participants) | 15 | 6
  Week 12 | 12.6 (24.22) | 4.7 (4.46)
  Week 13: number analyzed (Participants) | 11 | 5
  Week 13 | 5.8 (6.06) | 4.0 (3.81)
  Week 14: number analyzed (Participants) | 11 | 4
  Week 14 | 5.9 (7.30) | 2.5 (3.00)
  Week 15: number analyzed (Participants) | 11 | 3
  Week 15 | 4.9 (6.55) | 3.0 (5.20)
  Week 16: number analyzed (Participants) | 10 | 3
  Week 16 | 6.6 (8.35) | 2.3 (4.04)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 1: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.188, Negative binomial regression; LS Mean Difference = 1.70, 95% CI 2-sided [0.77 to 3.73], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 2: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.207, Negative binomial regression; LS Mean Difference = 1.81, 95% CI 2-sided [0.72 to 4.54], Standard Error of Mean 0.85
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 3: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.317, Negative binomial regression; LS Mean Difference = 1.71, 95% CI 2-sided [0.60 to 4.93], Standard Error of Mean 0.92
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 4: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.554, Negative binomial regression; LS Mean Difference = 1.36, 95% CI 2-sided [0.50 to 3.71], Standard Error of Mean 0.70
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 5: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.581, Negative binomial regression; LS Mean Difference = 0.78, 95% CI 2-sided [0.32 to 1.89], Standard Error of Mean 0.35
Statistical Analysis 6: Comparison: Tanezumab vs Placebo; Week 6: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.252, Negative binomial regression; LS Mean Difference = 0.61, 95% CI 2-sided [0.26 to 1.43], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Tanezumab vs Placebo; Week 7: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.365, Negative binomial regression; LS Mean Difference = 0.65, 95% CI 2-sided [0.26 to 1.64], Standard Error of Mean 0.31
Statistical Analysis 8: Comparison: Tanezumab vs Placebo; Week 8: Negative binomial regression model with model terms for treatment as a main effect. P-value was based on negative binomial regression model from pairwise comparisons. LS mean difference and corresponding 95% CI were estimated from the corresponding negative binomial regression model; Test type: Superiority or Other; p = 0.212, Negative binomial regression; LS Mean Difference = 0.58, 95% CI 2-sided [0.25 to 1.36], Standard Error of Mean 0.25

13. Secondary Outcome: Change From Baseline in Opioid-Related Symptom Distress Scale (OR-SDS) at Weeks 2, 4, 6, 12, and 16
Description: OR-SDS: participant-rated levels of frequency (F), severity (S), degree of bother (DoB) for 10 symptoms: fatigue, drowsiness, concentration, confusion, nausea, dizziness, constipation, itching, difficulty with urination, retching/vomiting. For each symptom levels of F, S and DoB scored as: frequency (0 to 4:'did not have' to 'almost constantly'), severity (0 to 4:'did not have' to 'very severe'), degree of bother (0 to 5:'did not have' to 'very much'). Mean of F, S and DoB was calculated for each symptom to derive composite scores/multi-domain average (MDA) scores which ranges from 0 to 4.33. Higher MDA=worse symptom. Composite scores for frequency (FCS), severity (SCS), degree of bother, and MDA were calculated as mean of these scores across 10 symptoms and had same ranges as individual scores frequency (0 to 4:'did not have' to 'almost constantly'), severity (0 to 4:'did not have' to 'very severe'), degree of bother (0 to 5:'did not have' to 'very much'); higher scores=more distress
Time Frame: Baseline, Week 2, 4, 6, 12, 16
Population: ITT population. Overall number of participants analyzed=participants who were evaluable for this measure; number analyzed=participants evaluable at specific time points; "0" in number analyzed field signifies no participant was evaluable for the parameter at this time point. For time points after Week 6 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 29
units on a scale
  Baseline Fatigue MDA: number analyzed (Participants) | 20 | 26
  Baseline Fatigue MDA | 2.05 (0.61) | 2.33 (0.53)
  Change at Week 2 Fatigue MDA: number analyzed (Participants) | 17 | 21
  Change at Week 2 Fatigue MDA | 0.1 (0.46) | -0.3 (0.56)
  Change at Week 4 Fatigue MDA: number analyzed (Participants) | 11 | 21
  Change at Week 4 Fatigue MDA | -0.2 (0.58) | -0.2 (0.57)
  Change at Week 6 Fatigue MDA: number analyzed (Participants) | 9 | 21
  Change at Week 6 Fatigue MDA | -0.3 (0.62) | -0.2 (0.43)
  Change at Week 12 Fatigue MDA: number analyzed (Participants) | 5 | 5
  Change at Week 12 Fatigue MDA | -0.3 (0.53) | -0.4 (0.76)
  Change at Week 16 Fatigue MDA: number analyzed (Participants) | 4 | 5
  Change at Week 16 Fatigue MDA | -0.5 (0.58) | -0.4 (0.15)
  Baseline Drowsiness MDA: number analyzed (Participants) | 15 | 23
  Baseline Drowsiness MDA | 1.89 (0.70) | 2.43 (0.81)
  Change at Week 2 Drowsiness MDA: number analyzed (Participants) | 12 | 17
  Change at Week 2 Drowsiness MDA | -0.1 (0.66) | -0.4 (0.84)
  Change at Week 4 Drowsiness MDA: number analyzed (Participants) | 10 | 17
  Change at Week 4 Drowsiness MDA | 0.1 (0.89) | -0.2 (0.65)
  Change at Week 6 Drowsiness MDA: number analyzed (Participants) | 8 | 14
  Change at Week 6 Drowsiness MDA | 0.0 (0.62) | -0.3 (0.76)
  Change at Week 12 Drowsiness MDA: number analyzed (Participants) | 7 | 6
  Change at Week 12 Drowsiness MDA | -0.3 (0.77) | -0.9 (0.96)
  Change at Week 16 Drowsiness MDA: number analyzed (Participants) | 4 | 4
  Change at Week 16 Drowsiness MDA | -0.6 (0.92) | -0.5 (0.64)
  Baseline Inability to concentrate (ITC) MDA: number analyzed (Participants) | 10 | 16
  Baseline Inability to concentrate (ITC) MDA | 1.53 (0.65) | 2.02 (0.51)
  Change at Week 2 ITC MDA: number analyzed (Participants) | 8 | 12
  Change at Week 2 ITC MDA | 0.2 (0.40) | -0.2 (0.46)
  Change at Week 4 ITC MDA: number analyzed (Participants) | 7 | 7
  Change at Week 4 ITC MDA | 0.1 (0.98) | -0.3 (0.23)
  Change at Week 6 ITC MDA: number analyzed (Participants) | 6 | 7
  Change at Week 6 ITC MDA | 0.2 (0.81) | -0.1 (0.38)
  Change at Week 12 ITC MDA: number analyzed (Participants) | 4 | 3
  Change at Week 12 ITC MDA | -0.2 (0.84) | -0.3 (0.33)
  Change at Week 16 ITC MDA: number analyzed (Participants) | 3 | 2
  Change at Week 16 ITC MDA | -0.1 (1.07) | -0.5 (0.24)
  Baseline Nausea MDA: number analyzed (Participants) | 11 | 8
  Baseline Nausea MDA | 2.18 (0.70) | 2.08 (0.87)
  Change at Week 2 Nausea MDA: number analyzed (Participants) | 8 | 6
  Change at Week 2 Nausea MDA | -0.0 (0.77) | 0.0 (0.67)
  Change at Week 4 Nausea MDA: number analyzed (Participants) | 6 | 3
  Change at Week 4 Nausea MDA | 0.1 (0.34) | -0.2 (0.38)
  Change at Week 6 Nausea MDA: number analyzed (Participants) | 3 | 3
  Change at Week 6 Nausea MDA | -0.7 (0.67) | 0.6 (0.77)
  Change at Week 12 Nausea MDA: number analyzed (Participants) | 0 | 0
  Change at Week 16 Nausea MDA: number analyzed (Participants) | 0 | 0
  Baseline Dizziness MDA: number analyzed (Participants) | 9 | 10
  Baseline Dizziness MDA | 1.70 (0.42) | 1.70 (0.48)
  Change at Week 2 Dizziness MDA: number analyzed (Participants) | 6 | 7
  Change at Week 2 Dizziness MDA | 0.5 (0.46) | 0.0 (0.36)
  Change at Week 4 Dizziness MDA: number analyzed (Participants) | 5 | 6
  Change at Week 4 Dizziness MDA | 0.5 (0.80) | -0.3 (0.37)
  Change at Week 6 Dizziness MDA: number analyzed (Participants) | 2 | 3
  Change at Week 6 Dizziness MDA | 0.5 (0.24) | -0.2 (0.38)
  Change at Week 12 Dizziness MDA: number analyzed (Participants) | 0 | 2
  Change at Week 12 Dizziness MDA |  | -0.3 (0.47)
  Change at Week 16 Dizziness MDA: number analyzed (Participants) | 0 | 3
  Change at Week 16 Dizziness MDA |  | -0.2 (0.51)
  Baseline Constipation MDA: number analyzed (Participants) | 19 | 15
  Baseline Constipation MDA | 1.96 (0.77) | 2.40 (1.02)
  Change at Week 2 Constipation MDA: number analyzed (Participants) | 10 | 11
  Change at Week 2 Constipation MDA | -0.1 (1.31) | 0.1 (1.32)
  Change at Week 4 Constipation MDA: number analyzed (Participants) | 7 | 10
  Change at Week 4 Constipation MDA | 0.5 (0.88) | -0.2 (0.67)
  Change at Week 6 Constipation MDA: number analyzed (Participants) | 5 | 10
  Change at Week 6 Constipation MDA | 0.5 (0.90) | 0.0 (0.52)
  Change at Week 12 Constipation MDA: number analyzed (Participants) | 5 | 4
  Change at Week 12 Constipation MDA | -0.2 (0.80) | -0.5 (1.73)
  Change at Week 16 Constipation MDA: number analyzed (Participants) | 2 | 1
  Change at Week 16 Constipation MDA | 1.2 (1.65) | 0.0
  Baseline Itching MDA: number analyzed (Participants) | 4 | 4
  Baseline Itching MDA | 1.83 (0.58) | 1.83 (0.33)
  Change at Week 2 Itching MDA: number analyzed (Participants) | 2 | 4
  Change at Week 2 Itching MDA | 0.0 (0.00) | -0.2 (0.33)
  Change at Week 4 Itching MDA: number analyzed (Participants) | 1 | 3
  Change at Week 4 Itching MDA | -1.0 | 0.2 (0.19)
  Change at Week 6 Itching MDA: number analyzed (Participants) | 2 | 2
  Change at Week 6 Itching MDA | -0.7 (0.94) | 0.3 (0.00)
  Change at Week 12 Itching MDA: number analyzed (Participants) | 0 | 0
  Change at Week 16 Itching MDA: number analyzed (Participants) | 0 | 0
  Baseline Difficulty with urination(DWU) MDA: number analyzed (Participants) | 4 | 5
  Baseline Difficulty with urination(DWU) MDA | 1.58 (0.50) | 2.27 (1.21)
  Change at Week 2 DWU MDA: number analyzed (Participants) | 4 | 4
  Change at Week 2 DWU MDA | 0.5 (0.79) | 0.0 (0.27)
  Change at Week 4 DWU MDA: number analyzed (Participants) | 4 | 1
  Change at Week 4 DWU MDA | 0.9 (1.10) | 0.0
  Change at Week 6 DWU MDA: number analyzed (Participants) | 2 | 2
  Change at Week 6 DWU MDA | 0.3 (0.94) | -0.8 (0.24)
  Change at Week 12 DWU MDA: number analyzed (Participants) | 1 | 1
  Change at Week 12 DWU MDA | -0.3 | 0.0
  Change at Week 16 DWU MDA: number analyzed (Participants) | 0 | 1
  Change at Week 16 DWU MDA |  | -0.7
  Baseline Confusion MDA: number analyzed (Participants) | 1 | 7
  Baseline Confusion MDA | 1.67 | 1.67 (0.38)
  Change at Week 2 Confusion MDA: number analyzed (Participants) | 1 | 3
  Change at Week 2 Confusion MDA | -0.7 | -0.4 (0.51)
  Change at Week 4 Confusion MDA: number analyzed (Participants) | 1 | 3
  Change at Week 4 Confusion MDA | -0.7 | -0.2 (0.38)
  Change at Week 6 Confusion MDA: number analyzed (Participants) | 1 | 2
  Change at Week 6 Confusion MDA | -0.7 | 0.3 (0.47)
  Change at Week 12 Confusion MDA: number analyzed (Participants) | 1 | 0
  Change at Week 12 Confusion MDA | -0.7 |
  Change at Week 16 Confusion MDA: number analyzed (Participants) | 0 | 1
  Change at Week 16 Confusion MDA |  | 0.3
  Baseline Retching/Vomiting MDA: number analyzed (Participants) | 3 | 6
  Baseline Retching/Vomiting MDA | 2.56 (0.69) | 2.06 (0.61)
  Change at Week 2 Retching/Vomiting MDA: number analyzed (Participants) | 2 | 3
  Change at Week 2 Retching/Vomiting MDA | 0.2 (0.24) | -0.7 (0.33)
  Change at Week 4 Retching/Vomiting MDA: number analyzed (Participants) | 2 | 3
  Change at Week 4 Retching/Vomiting MDA | -0.7 (0.47) | 0.0 (0.33)
  Change at Week 6 Retching/Vomiting MDA: number analyzed (Participants) | 1 | 2
  Change at Week 6 Retching/Vomiting MDA | -0.3 | 0.7 (0.94)
  Change at Week 12 Retching/Vomiting MDA: number analyzed (Participants) | 0 | 0
  Change at Week 16 Retching/Vomiting MDA: number analyzed (Participants) | 0 | 0
  Baseline Frequency Composite Score (FCS) | 1.82 (0.52) | 2.14 (0.73)
  Change at Week 2 FCS: number analyzed (Participants) | 25 | 27
  Change at Week 2 FCS | -0.0 (0.55) | -0.2 (0.66)
  Change at Week 4 FCS: number analyzed (Participants) | 21 | 24
  Change at Week 4 FCS | -0.0 (0.76) | -0.0 (0.69)
  Change at Week 6 FCS: number analyzed (Participants) | 16 | 22
  Change at Week 6 FCS | -0.3 (0.55) | -0.1 (0.48)
  Change at Week 12 FCS: number analyzed (Participants) | 10 | 7
  Change at Week 12 FCS | -0.3 (0.48) | -0.4 (0.55)
  Change at Week 16 FCS: number analyzed (Participants) | 6 | 5
  Change at Week 16 FCS | -0.2 (0.88) | -0.2 (0.46)
  Baseline Severity Composite Score (SCS) | 1.60 (0.50) | 1.78 (0.42)
  Change at Week 2 SCS: number analyzed (Participants) | 25 | 26
  Change at Week 2 SCS | 0.0 (0.53) | 0.0 (0.51)
  Change at Week 4 SCS: number analyzed (Participants) | 21 | 24
  Change at Week 4 SCS | 0.1 (0.62) | -0.1 (0.50)
  Change at Week 6 SCS: number analyzed (Participants) | 16 | 22
  Change at Week 6 SCS | -0.0 (0.44) | -0.1 (0.44)
  Change at Week 12 SCS: number analyzed (Participants) | 10 | 7
  Change at Week 12 SCS | 0.0 (0.31) | -0.3 (0.52)
  Change at Week 16 SCS: number analyzed (Participants) | 6 | 5
  Change at Week 16 SCS | 0.0 (0.97) | -0.1 (0.24)
  Baseline Bother Composite Score | 2.29 (0.74) | 2.49 (0.73)
  Change at Week 2 Bother Composite Score: number analyzed (Participants) | 25 | 26
  Change at Week 2 Bother Composite Score | -0.0 (0.61) | -0.1 (0.70)
  Change at Week 4 Bother Composite Score: number analyzed (Participants) | 21 | 24
  Change at Week 4 Bother Composite Score | -0.0 (0.79) | -0.1 (0.85)
  Change at Week 6 Bother Composite Score: number analyzed (Participants) | 16 | 22
  Change at Week 6 Bother Composite Score | -0.1 (0.62) | -0.2 (0.59)
  Change at Week 12 Bother Composite Score: number analyzed (Participants) | 10 | 7
  Change at Week 12 Bother Composite Score | -0.1 (1.05) | -0.5 (0.85)
  Change at Week 16 Bother Composite Score: number analyzed (Participants) | 6 | 5
  Change at Week 16 Bother Composite Score | -0.4 (1.13) | -0.6 (0.84)
  Baseline MDA Composite Score | 1.90 (0.49) | 2.14 (0.53)
  Change at Week 2 MDA Composite Score: number analyzed (Participants) | 25 | 27
  Change at Week 2 MDA Composite Score | -0.0 (0.46) | -0.1 (0.51)
  Change at Week 4 MDA Composite Score: number analyzed (Participants) | 21 | 24
  Change at Week 4 MDA Composite Score | 0.0 (0.62) | -0.1 (0.61)
  Change at Week 6 MDA Composite Score: number analyzed (Participants) | 16 | 22
  Change at Week 6 MDA Composite Score | -0.1 (0.42) | -0.1 (0.41)
  Change at Week 12 MDA Composite Score: number analyzed (Participants) | 10 | 7
  Change at Week 12 MDA Composite Score | -0.1 (0.57) | -0.4 (0.50)
  Change at Week 16 MDA Composite Score: number analyzed (Participants) | 6 | 5
  Change at Week 16 MDA Composite Score | -0.2 (0.88) | -0.3 (0.25)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 2 (Fatigue MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.215, ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [-0.13 to 0.55], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Change at Week 4 (Fatigue MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.947, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.45 to 0.42], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Change at Week 6 (Fatigue MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.341, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.56 to 0.20], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 2 (Drowsiness MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.180, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-0.83 to 0.17], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Change at Week 4 (Drowsiness MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.509, ANCOVA; LS Mean Difference = 0.20, 95% CI 2-sided [-0.43 to 0.84], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Tanezumab vs Placebo; Change at Week 6 (Drowsiness MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.767, ANCOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-0.62 to 0.82], Standard Error of Mean 0.34
Statistical Analysis 7: Comparison: Tanezumab vs Placebo; Change at Week 2 (Inability to Concentrate MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.108, ANCOVA; LS Mean Difference = 0.42, 95% CI 2-sided [-0.11 to 0.95], Standard Error of Mean 0.25
Statistical Analysis 8: Comparison: Tanezumab vs Placebo; Change at Week 4 (Inability to Concentrate MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.280, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-1.26 to 0.41], Standard Error of Mean 0.37
Statistical Analysis 9: Comparison: Tanezumab vs Placebo; Change at Week 6 (Inability to Concentrate MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.747, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-1.53 to 1.15], Standard Error of Mean 0.57
Statistical Analysis 10: Comparison: Tanezumab vs Placebo; Change at Week 2 (Nausea MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.991, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.87 to 0.88], Standard Error of Mean 0.39
Statistical Analysis 11: Comparison: Tanezumab vs Placebo; Change at Week 4 (Nausea MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.335, ANCOVA; LS Mean Difference = 0.29, 95% CI 2-sided [-0.41 to 0.99], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Tanezumab vs Placebo; Change at Week 6 (Nausea MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.159, ANCOVA; LS Mean Difference = -1.55, 95% CI 2-sided [-4.57 to 1.48], Standard Error of Mean 0.70
Statistical Analysis 13: Comparison: Tanezumab vs Placebo; Change at Week 2 (Dizziness MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.136, ANCOVA; LS Mean Difference = 0.39, 95% CI 2-sided [-0.16 to 0.94], Standard Error of Mean 0.23
Statistical Analysis 14: Comparison: Tanezumab vs Placebo; Change at Week 6 (Dizziness MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.186, ANCOVA; LS Mean Difference = 1.22, 95% CI 2-sided [-3.46 to 5.90], Standard Error of Mean 0.37
Statistical Analysis 15: Comparison: Tanezumab vs Placebo; Change at Week 2 (Constipation MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.292, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-1.52 to 0.49], Standard Error of Mean 0.48
Statistical Analysis 16: Comparison: Tanezumab vs Placebo; Change at Week 4 (Constipation MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.225, ANCOVA; LS Mean Difference = 0.48, 95% CI 2-sided [-0.34 to 1.30], Standard Error of Mean 0.38
Statistical Analysis 17: Comparison: Tanezumab vs Placebo; Change at Week 6 (Constipation MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.517, ANCOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.58 to 1.07], Standard Error of Mean 0.36
Statistical Analysis 18: Comparison: Tanezumab vs Placebo; Change at Week 2 (Itching MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 1.000, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-2.48 to 2.48], Standard Error of Mean 0.58
Statistical Analysis 19: Comparison: Tanezumab vs Placebo; Change at Week 4 (Itching MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.00, 95% CI 2-sided [-1.01 to -0.99], Standard Error of Mean 0.00
Statistical Analysis 20: Comparison: Tanezumab vs Placebo; Change at Week 2 (Difficulty with Urination MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.362, ANCOVA; LS Mean Difference = 0.44, 95% CI 2-sided [-0.75 to 1.63], Standard Error of Mean 0.43
Statistical Analysis 21: Comparison: Tanezumab vs Placebo; Change at Week 4 (Difficulty with Urination MDA): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 1.000, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-51.87 to 51.87], Standard Error of Mean 4.08
Statistical Analysis 22: Comparison: Tanezumab vs Placebo; Change at Week 4 (Retching/Vomiting MDR): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.031, ANCOVA; LS Mean Difference = -2.03, 95% CI 2-sided [-3.30 to -0.76], Standard Error of Mean 0.10
Statistical Analysis 23: Comparison: Tanezumab vs Placebo; Change at Week 2 (Frequency Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.886, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.28 to 0.32], Standard Error of Mean 0.15
Statistical Analysis 24: Comparison: Tanezumab vs Placebo; Change at Week 4 (Frequency Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.660, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.52 to 0.33], Standard Error of Mean 0.21
Statistical Analysis 25: Comparison: Tanezumab vs Placebo; Change at Week 6 (Frequency Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.238, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.54 to 0.14], Standard Error of Mean 0.17
Statistical Analysis 26: Comparison: Tanezumab vs Placebo; Change at Week 2 (Severity Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.360, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.42 to 0.16], Standard Error of Mean 0.14
Statistical Analysis 27: Comparison: Tanezumab vs Placebo; Change at Week 4 (Severity Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.278, ANCOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-0.16 to 0.54], Standard Error of Mean 0.17
Statistical Analysis 28: Comparison: Tanezumab vs Placebo; Change at Week 6 (Severity Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.809, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.34 to 0.27], Standard Error of Mean 0.15
Statistical Analysis 29: Comparison: Tanezumab vs Placebo; Change at Week 2 (Bother Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.944, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.35 to 0.38], Standard Error of Mean 0.18
Statistical Analysis 30: Comparison: Tanezumab vs Placebo; Change at Week 4 (Bother Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.892, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.48 to 0.55], Standard Error of Mean 0.26
Statistical Analysis 31: Comparison: Tanezumab vs Placebo; Change at Week 6 (Bother Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.884, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.39 to 0.45], Standard Error of Mean 0.21
Statistical Analysis 32: Comparison: Tanezumab vs Placebo; Change at Week 2 (MDA Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.919, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.26 to 0.28], Standard Error of Mean 0.13
Statistical Analysis 33: Comparison: Tanezumab vs Placebo; Change at Week 4 (MDA Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.752, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.33 to 0.45], Standard Error of Mean 0.19
Statistical Analysis 34: Comparison: Tanezumab vs Placebo; Change at Week 6 (MDA Composite Score): LS mean difference and corresponding 95% CI were estimated from the corresponding repeated measures ANCOVA model; Test type: Superiority or Other; p = 0.715, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.34 to 0.24], Standard Error of Mean 0.14

14. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Pain Interference With Function Composite Score and Individual Pain Interference Item Scores of General Activity, Walking Ability and Normal Work at Weeks 1, 2, 4, 6, 8, 12, and 16: BOCF
Description: Participant-rated 11 point Likert rating scale ranging from 0 (does not interfere) to 10 (completely interferes) assessed interference of pain in functional activities (general activity, walking ability, and normal work) in past 24 hours. Measures were scored by individual item as well as function composite score (calculated by taking mean of individual interference scores), both (individual scores and composite scores) ranging from 0 to 10 with lower scores being indicative of less pain interference.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Here "overall number of participants analyzed" signifies those participants who were evaluable for this measure. For time points after Week 8 inferential statistics were not performed because post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 27
units on a scale
  Baseline Composite Score | 4.90 (1.56) | 5.19 (1.66)
  Change at Week 1 Composite Score | -0.3 (1.49) | -0.8 (2.17)
  Change at Week 2 Composite Score | -0.9 (1.41) | -1.1 (1.98)
  Change at Week 4 Composite Score | -1.3 (1.56) | -1.2 (1.83)
  Change at Week 6 Composite Score | -1.1 (1.53) | -0.9 (1.98)
  Change at Week 8 Composite Score | -1.0 (1.92) | -0.8 (1.98)
  Change at Week 12 Composite Score | -0.8 (1.56) | -0.1 (0.89)
  Change at Week 16 Composite Score | -0.9 (1.50) | -0.2 (0.80)
  Baseline General Activity | 5.41 (1.34) | 5.41 (1.47)
  Change at Week 1 General Activity | -0.5 (1.74) | -0.8 (2.06)
  Change at Week 2 General Activity | -1.0 (1.80) | -0.9 (2.27)
  Change at Week 4 General Activity | -1.4 (2.04) | -1.3 (1.95)
  Change at Week 6 General Activity | -1.1 (1.79) | -0.9 (2.15)
  Change at Week 8 General Activity | -1.1 (2.13) | -0.8 (2.40)
  Change at Week 12 General Activity | -0.7 (2.03) | -0.1 (1.53)
  Change at Week 16 General Activity | -1.0 (1.66) | -0.3 (1.24)
  Baseline Walking Ability | 4.4 (2.32) | 5.5 (2.04)
  Change at Week 1 Walking Ability | -0.0 (1.99) | -0.7 (2.65)
  Change at Week 2 Walking Ability | -0.1 (2.20) | -0.5 (2.32)
  Change at Week 4 Walking Ability | -0.7 (1.92) | -0.9 (2.48)
  Change at Week 6 Walking Ability | -0.6 (2.00) | -0.8 (2.34)
  Change at Week 8 Walking Ability | -0.5 (2.46) | -0.5 (2.16)
  Change at Week 12 Walking Ability | -0.5 (2.03) | 0.0 (1.23)
  Change at Week 16 Walking Ability | -0.7 (1.98) | -0.2 (0.80)
  Baseline Normal Work | 5.19 (1.92) | 5.69 (2.26)
  Change at Week 1 Normal Work | -0.37 (2.37) | -0.42 (2.76)
  Change at Week 2 Normal Work | -1.04 (1.87) | -0.65 (2.97)
  Change at Week 4 Normal Work | -1.15 (2.09) | -1.23 (2.52)
  Change at Week 6 Normal Work | -0.74 (2.35) | -0.69 (2.72)
  Change at Week 8 Normal Work | -0.85 (2.18) | -0.65 (2.17)
  Change at Week 12 Normal Work | -0.67 (1.71) | 0.08 (1.44)
  Change at Week 16 Normal Work | -0.70 (1.75) | -0.19 (0.94)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 1 (Composite Score): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.666, ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [-0.77 to 1.18], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Change at Week 2 (Composite Score): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.745, ANCOVA; LS Mean Difference = 0.16, 95% CI 2-sided [-0.86 to 1.18], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Change at Week 4 (Composite Score): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.749, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-1.14 to 0.83], Standard Error of Mean 0.48
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 6 (Composite Score): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.794, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-1.16 to 0.90], Standard Error of Mean 0.50
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Change at Week 8 (Composite Score): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.772, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-1.33 to 1.00], Standard Error of Mean 0.56
Statistical Analysis 6: Comparison: Tanezumab vs Placebo; Change at Week 1 (General Activity): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.547, ANCOVA; LS Mean Difference = 0.31, 95% CI 2-sided [-0.73 to 1.34], Standard Error of Mean 0.50
Statistical Analysis 7: Comparison: Tanezumab vs Placebo; Change at Week 2 (General Activity): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.650, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-1.43 to 0.91], Standard Error of Mean 0.57
Statistical Analysis 8: Comparison: Tanezumab vs Placebo; Change at Week 4 (General Activity): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.808, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-1.27 to 1.00], Standard Error of Mean 0.55
Statistical Analysis 9: Comparison: Tanezumab vs Placebo; Change at Week 6 (General Activity): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.915, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-1.19 to 1.07], Standard Error of Mean 0.55
Statistical Analysis 10: Comparison: Tanezumab vs Placebo; Change at Week 8 (General Activity): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.757, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-1.54 to 1.14], Standard Error of Mean 0.65
Statistical Analysis 11: Comparison: Tanezumab vs Placebo; Change at Week 1 (Walking Ability): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.987, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-1.19 to 1.17], Standard Error of Mean 0.57
Statistical Analysis 12: Comparison: Tanezumab vs Placebo; Change at Week 2 (Walking Ability): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.781, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-1.14 to 1.51], Standard Error of Mean 0.64
Statistical Analysis 13: Comparison: Tanezumab vs Placebo; Change at Week 4 (Walking Ability): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.834, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-1.13 to 1.38], Standard Error of Mean 0.61
Statistical Analysis 14: Comparison: Tanezumab vs Placebo; Change at Week 6 (Walking Ability): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.851, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-1.32 to 1.10], Standard Error of Mean 0.59
Statistical Analysis 15: Comparison: Tanezumab vs Placebo; Change at Week 8 (Walking Ability): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.701, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-1.68 to 1.15], Standard Error of Mean 0.68
Statistical Analysis 16: Comparison: Tanezumab vs Placebo; Change at Week 1 (Normal Work): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.453, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-1.68 to 0.77], Standard Error of Mean 0.59
Statistical Analysis 17: Comparison: Tanezumab vs Placebo; Change at Week 2 (Normal Work): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.258, ANCOVA; LS Mean Difference = -0.77, 95% CI 2-sided [-2.15 to 0.60], Standard Error of Mean 0.67
Statistical Analysis 18: Comparison: Tanezumab vs Placebo; Change at Week 4 (Normal Work): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.736, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-1.53 to 1.09], Standard Error of Mean 0.64
Statistical Analysis 19: Comparison: Tanezumab vs Placebo; Change at Week 6 (Normal Work): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.491, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-1.76 to 0.87], Standard Error of Mean 0.64
Statistical Analysis 20: Comparison: Tanezumab vs Placebo; Change at Week 8 (Normal Work): ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.695, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-1.53 to 1.04], Standard Error of Mean 0.62

15. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Pain Interference With Function Composite Score and Individual Pain Interference Item Scores at Weeks 1, 2, 4, 6, 8, 12, and 16: LOCF
Description: Participant-rated 11 point Likert rating scale ranging from 0 (does not interfere) to 10 (completely interferes) assessed interference of pain in functional activities (general activity, walking ability, and normal work) in past 24 hours. Measures were scored by individual item as well as function composite score (calculated by taking mean of individual interference scores), both (individual items and composite scores) ranging from 0 to 10 with lower scores being indicative of less pain interference.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 27
units on a scale
  Baseline Composite Score: number analyzed (Participants) | 27 | 26
  Baseline Composite Score | 4.90 (1.56) | 5.19 (1.66)
  Change at Week 1 Composite Score: number analyzed (Participants) | 20 | 21
  Change at Week 1 Composite Score | -0.4 (1.73) | -0.9 (2.39)
  Change at Week 2 Composite Score: number analyzed (Participants) | 24 | 25
  Change at Week 2 Composite Score | -1.0 (1.47) | -1.5 (2.42)
  Change at Week 4 Composite Score: number analyzed (Participants) | 25 | 25
  Change at Week 4 Composite Score | -1.4 (1.57) | -1.2 (2.01)
  Change at Week 6 Composite Score: number analyzed (Participants) | 25 | 25
  Change at Week 6 Composite Score | -1.3 (1.64) | -1.0 (2.13)
  Change at Week 8 Composite Score: number analyzed (Participants) | 25 | 25
  Change at Week 8 Composite Score | -1.3 (1.96) | -0.8 (2.13)
  Change at Week 12 Composite Score: number analyzed (Participants) | 25 | 25
  Change at Week 12 Composite Score | -1.3 (2.10) | -0.9 (1.94)
  Change at Week 16 Composite Score: number analyzed (Participants) | 25 | 25
  Change at Week 16 Composite Score | -1.3 (2.11) | -0.9 (1.92)
  Baseline General Activity | 5.41 (1.34) | 5.41 (1.47)
  Change at Week 1 General Activity: number analyzed (Participants) | 20 | 21
  Change at Week 1 General Activity | -0.7 (2.01) | -1.0 (2.29)
  Change at Week 2 General Activity: number analyzed (Participants) | 24 | 25
  Change at Week 2 General Activity | -1.1 (1.91) | -1.2 (2.73)
  Change at Week 4 General Activity: number analyzed (Participants) | 25 | 26
  Change at Week 4 General Activity | -1.5 (2.08) | -1.0 (2.46)
  Change at Week 6 General Activity: number analyzed (Participants) | 25 | 26
  Change at Week 6 General Activity | -1.4 (2.08) | -0.8 (2.61)
  Change at Week 8 General Activity: number analyzed (Participants) | 25 | 26
  Change at Week 8 General Activity | -1.4 (2.31) | -0.5 (2.87)
  Change at Week 12 General Activity: number analyzed (Participants) | 25 | 26
  Change at Week 12 General Activity | -1.2 (2.55) | -0.6 (2.80)
  Change at Week 16 General Activity: number analyzed (Participants) | 25 | 26
  Change at Week 16 General Activity | -1.4 (2.47) | -0.7 (2.76)
  Baseline Walking Ability: number analyzed (Participants) | 27 | 26
  Baseline Walking Ability | 4.4 (2.32) | 5.5 (2.04)
  Change at Week 1 Walking Ability: number analyzed (Participants) | 20 | 21
  Change at Week 1 Walking Ability | -0.1 (2.33) | -0.8 (2.94)
  Change at Week 2 Walking Ability: number analyzed (Participants) | 24 | 25
  Change at Week 2 Walking Ability | -0.2 (2.33) | -1.0 (2.89)
  Change at Week 4 Walking Ability: number analyzed (Participants) | 25 | 25
  Change at Week 4 Walking Ability | -0.8 (1.98) | -0.9 (2.64)
  Change at Week 6 Walking Ability: number analyzed (Participants) | 25 | 25
  Change at Week 6 Walking Ability | -0.6 (2.31) | -1.0 (2.52)
  Change at Week 8 Walking Ability: number analyzed (Participants) | 25 | 25
  Change at Week 8 Walking Ability | -0.8 (2.66) | -0.5 (2.43)
  Change at Week 12 Walking Ability: number analyzed (Participants) | 25 | 25
  Change at Week 12 Walking Ability | -0.5 (2.69) | -0.4 (2.31)
  Change at Week 16 Walking Ability: number analyzed (Participants) | 25 | 25
  Change at Week 16 Walking Ability | -0.5 (2.76) | -0.4 (2.36)
  Baseline Normal Work: number analyzed (Participants) | 27 | 26
  Baseline Normal Work | 5.19 (1.92) | 5.69 (2.26)
  Change at Week 1 Normal Work: number analyzed (Participants) | 20 | 21
  Change at Week 1 Normal Work | -0.50 (2.76) | -0.52 (3.08)
  Change at Week 2 Normal Work: number analyzed (Participants) | 24 | 25
  Change at Week 2 Normal Work | -1.04 (2.12) | -1.00 (3.46)
  Change at Week 4 Normal Work: number analyzed (Participants) | 25 | 25
  Change at Week 4 Normal Work | -1.24 (2.15) | -1.16 (2.69)
  Change at Week 6 Normal Work: number analyzed (Participants) | 25 | 25
  Change at Week 6 Normal Work | -1.04 (2.62) | -0.72 (2.91)
  Change at Week 8 Normal Work: number analyzed (Participants) | 25 | 25
  Change at Week 8 Normal Work | -1.08 (2.53) | -0.84 (2.39)
  Change at Week 12 Normal Work: number analyzed (Participants) | 25 | 25
  Change at Week 12 Normal Work | -1.36 (2.41) | -0.64 (2.45)
  Change at Week 16 Normal Work: number analyzed (Participants) | 25 | 25
  Change at Week 16 Normal Work | -1.52 (2.40) | -0.68 (2.44)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.897, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-1.34 to 1.19], Standard Error of Mean 0.60
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.643, ANCOVA; LS Mean Difference = 0.26, 95% CI 2-sided [-0.90 to 1.43], Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; p = 0.464, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-1.45 to 0.68], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority or Other; p = 0.593, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-1.46 to 0.86], Standard Error of Mean 0.56
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 5]; Test type: Superiority or Other; p = 0.423, ANCOVA; LS Mean Difference = -0.50, 95% CI 2-sided [-1.77 to 0.77], Standard Error of Mean 0.61
Statistical Analysis 6: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 6]; Test type: Superiority or Other; p = 0.805, ANCOVA; LS Mean Difference = 0.16, 95% CI 2-sided [-1.21 to 1.54], Standard Error of Mean 0.65
Statistical Analysis 7: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.882, ANCOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-1.30 to 1.51], Standard Error of Mean 0.68
Statistical Analysis 8: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 8]; Test type: Superiority or Other; p = 0.446, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-1.79 to 0.81], Standard Error of Mean 0.63
Statistical Analysis 9: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 9]; Test type: Superiority or Other; p = 0.604, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-1.77 to 1.05], Standard Error of Mean 0.68
Statistical Analysis 10: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 10]; Test type: Superiority or Other; p = 0.393, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-2.24 to 0.91], Standard Error of Mean 0.76
Statistical Analysis 11: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 11]; Test type: Superiority or Other; p = 0.399, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-2.33 to 0.97], Standard Error of Mean 0.79
Statistical Analysis 12: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p = 0.876, ANCOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-1.43 to 1.66], Standard Error of Mean 0.75
Statistical Analysis 13: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.740, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-1.58 to 1.14], Standard Error of Mean 0.66
Statistical Analysis 14: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 14]; Test type: Superiority or Other; p = 0.854, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-1.56 to 1.31], Standard Error of Mean 0.69
Statistical Analysis 15: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 15]; Test type: Superiority or Other; p = 0.436, ANCOVA; LS Mean Difference = -0.62, 95% CI 2-sided [-2.24 to 1.00], Standard Error of Mean 0.78
Statistical Analysis 16: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 16]; Test type: Superiority or Other; p = 0.087, ANCOVA; LS Mean Difference = -1.30, 95% CI 2-sided [-2.81 to 0.21], Standard Error of Mean 0.72
Statistical Analysis 17: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 17]; Test type: Superiority or Other; p = 0.278, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-2.40 to 0.72], Standard Error of Mean 0.75
Statistical Analysis 18: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 18]; Test type: Superiority or Other; p = 0.548, ANCOVA; LS Mean Difference = -0.42, 95% CI 2-sided [-1.84 to 1.00], Standard Error of Mean 0.69
Statistical Analysis 19: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.318, ANCOVA; LS Mean Difference = -0.77, 95% CI 2-sided [-2.33 to 0.79], Standard Error of Mean 0.75
Statistical Analysis 20: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 14, analysis 20]; Test type: Superiority or Other; p = 0.484, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-2.02 to 0.99], Standard Error of Mean 0.73

16. Secondary Outcome: Patient's Global Evaluation of Study Medication
Description: The Patient's Global Evaluation of Study Medication (PGESM) was a single item that assessed the participant's perception of his/her response to the study medication. It was a self-administered question that utilizes a 4-point Likert scale from 1="Poor" to 4="Excellent", where higher score represented better outcome.
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 29
units on a scale
  Week 1: number analyzed (Participants) | 21 | 24
  Week 1 | 2.7 (0.91) | 2.3 (0.81)
  Week 2: number analyzed (Participants) | 25 | 26
  Week 2 | 2.6 (0.82) | 2.4 (0.94)
  Week 4 | 2.4 (0.64) | 2.3 (0.90)
  Week 6 | 2.5 (0.75) | 2.3 (0.90)
  Week 8 | 2.7 (0.83) | 2.2 (0.86)
  Week 12 | 2.5 (0.75) | 2.3 (0.89)
  Week 16 | 2.6 (0.80) | 2.4 (0.94)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 1: P-value was calculated by Cochran-Mantel-Haenszel (CMH test) stratified by center; Test type: Superiority or Other; p = 0.399, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 2: P-value was calculated by CMH test stratified by center; Test type: Superiority or Other; p = 0.779, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 4: P-value was calculated by CMH test stratified by center; Test type: Superiority or Other; p = 0.922, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 6: P-value was calculated by CMH test stratified by center; Test type: Superiority or Other; p = 0.811, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 8: P-value was calculated by CMH test stratified by center; Test type: Superiority or Other; p = 0.237, Cochran-Mantel-Haenszel

17. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease (Cancer Pain) Activity at Weeks 1, 2, 4, 6, 8, 12, and 16: BOCF
Description: The Patient's Global Assessment of Cancer Pain was a global evaluation that utilized a 5-point Likert scale with a score of 1 being the best (Very Good) and a score of 5 being the worst (Very Poor), where higher score represented more pain.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Missing data were imputed using BOCF method. Here "overall number of participants analyzed" signifies participants evaluable for this measure. For time points after Week 8 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 26
units on a scale
  Baseline | 3.26 (0.66) | 2.92 (0.56)
  Change at Week 1 | -0.3 (0.62) | 0.2 (0.94)
  Change at Week 2 | -0.4 (0.57) | 0.0 (0.85)
  Change at Week 4 | -0.5 (0.75) | -0.2 (0.86)
  Change at Week 6 | -0.4 (0.80) | -0.3 (0.92)
  Change at Week 8 | -0.3 (0.91) | -0.1 (1.02)
  Change at Week 12 | -0.4 (0.63) | -0.1 (0.48)
  Change at Week 16 | -0.2 (0.51) | -0.0 (0.34)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 1: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.108, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.82 to 0.09], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Change at Week 2: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.202, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.70 to 0.16], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Change at Week 4: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.571, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.54 to 0.30], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 6: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.808, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.55 to 0.43], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Change at Week 8: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.913, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.57 to 0.51], Standard Error of Mean 0.26

18. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease (Cancer Pain) Activity at Weeks 1, 2, 4, 6, 8, 12, and 16: LOCF
Description: as for outcome 17
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Missing values were imputed using LOCF method. Here "overall number of participants analyzed" signifies participants who were evaluable for this measure. For time points after Week 8 inferential statistics were not done as post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 26
units on a scale
  Baseline | 3.26 (0.66) | 2.92 (0.56)
  Change at Week 1 | -0.3 (0.62) | 0.2 (0.94)
  Change at Week 2 | -0.4 (0.58) | -0.0 (0.96)
  Change at Week 4 | -0.5 (0.75) | -0.1 (1.07)
  Change at Week 6 | -0.5 (0.85) | -0.2 (1.13)
  Change at Week 8 | -0.4 (1.01) | 0.0 (1.20)
  Change at Week 12 | -0.4 (0.84) | -0.1 (1.14)
  Change at Week 16 | -0.3 (0.78) | -0.1 (1.13)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 1: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.108, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.82 to 0.09], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Change at Week 2: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.339, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.65 to 0.23], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Change at Week 4: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.408, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.67 to 0.28], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 6: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.686, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.67 to 0.45], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Change at Week 8: ANCOVA model included treatment and cancer type as fixed effects, baseline value as a covariate and study site as a random effect. LS mean difference and corresponding 95% CI were estimated from the corresponding ANCOVA model; Test type: Superiority or Other; p = 0.493, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.81 to 0.40], Standard Error of Mean 0.30

19. Secondary Outcome: Percentage of Participants Achieving Improvement of >=2 Points in Patient's Global Assessment Of Disease (Cancer Pain) Activity: BOCF
Description: as for outcome 17
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population. Missing values were imputed using BOCF method. Here "overall number of participants analyzed" signifies participants who were evaluable for this measure. Data was not summarized statistically at Week 12 and 16 because post Week 8 participants were eligible to roll-over into extension study A4091029 (NCT00830180).
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 26
percentage of participants
  Week 1 | 3.7 | 3.8
  Week 2 | 0 | 3.8
  Week 4 | 7.4 | 3.8
  Week 6 | 14.8 | 7.7
  Week 8 | 11.1 | 3.8
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 1: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.724, Fisher Exact; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.03 to 12.27]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 2: P-value was calculated using Fisher Extract method; Test type: Superiority or Other; p = 0.947, Fisher Exact
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 4: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.634, Fisher Exact; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.03 to 8.71]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 6: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.975, Fisher Exact; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.14 to 7.74]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 8: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.759, Fisher Exact; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.12 to 18.86]

20. Secondary Outcome: Percentage of Participants Achieving Improvement Of >=2 Points in Patient's Global Assessment Of Disease (Cancer Pain) Activity: LOCF
Description: as for outcome 17
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 26
percentage of participants
  Week 1 | 3.7 | 3.8
  Week 2 | 0 | 7.7
  Week 4 | 7.4 | 3.8
  Week 6 | 14.8 | 7.7
  Week 8 | 14.8 | 3.8
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 1: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.724, Fisher Exact; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.03 to 12.27]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 2: P-value was calculated using Fisher Extract test; Test type: Superiority or Other; p = 0.950, Fisher Exact
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 4: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.634, Fisher Exact; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.03 to 8.71]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 6: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.975, Fisher Exact; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.14 to 7.74]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 8: The odds ratio with 95% 2-sided CI for the treatment contrast was given; Test type: Superiority or Other; p = 0.578, Fisher Exact; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.17 to 23.89]

21. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 113 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 113 days
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo).
Measure: Number; unit: participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
participants
  AEs | 18 | 18
  SAEs | 7 | 4

22. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: Physical examinations included general appearance (skin, neck, eyes, ears, nose, throat), cardiovascular system (including rhythm and presence of other cardiac abnormalities, such as gallops, murmurs, and cardiomegaly), respiratory system, gastrointestinal system, genitourinary system, musculoskeletal system, and any additional assessments necessary to establish baseline status or evaluate symptoms or adverse experiences. Abnormalities in physical examination was based on investigator's discretion.
Time Frame: Baseline up to Week 16 or Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 23 | 28
Participants | 2 | 8

23. Secondary Outcome: Number of Participants With Abnormal Neurological Examination
Description: Neurological examinations assessed strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index finger and great toes in order to complete the neuropathy impairment score (NIS). NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items, from both the left and right side, where 24 items scored from 0 (normal) to 4 (paralysis) for muscle strength, higher score indicated higher abnormality/impairment, and 13 items scored from 0 (normal), 1 (decreased) and 2 (absent) for sensation, higher score indicated higher impairment. NIS possible overall score ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased impairment.
Time Frame: Week 2, 4, 6, 12, 16, Early Termination (up to 113 days)
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
participants
  Week 2 | 1 | 3
  Week 4 | 2 | 3
  Week 6 | 1 | 5
  Week 12 | 1 | 1
  Week 16 | 0 | 1
  Early Termination | 3 | 4

24. Secondary Outcome: Vital Sign Examination: Body Temperature
Time Frame: Baseline (Day 1 0H), Week 2, 4, 6, 12, 16, Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here N (number of participants analyzed) signifies the participants who were evaluable for this measure. n=participants evaluable at specific time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
degrees Celsius
  Baseline | 36.7 (0.18) | 36.6 (0.25)
  Week 2: number analyzed (Participants) | 27 | 27
  Week 2 | 36.7 (0.19) | 36.6 (0.27)
  Week 4: number analyzed (Participants) | 27 | 27
  Week 4 | 36.7 (0.18) | 36.6 (0.21)
  Week 6: number analyzed (Participants) | 23 | 25
  Week 6 | 36.6 (0.24) | 36.7 (0.26)
  Week 12: number analyzed (Participants) | 13 | 7
  Week 12 | 36.7 (0.18) | 36.6 (0.14)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 36.6 (0.16) | 36.7 (0.15)
  Early Termination: number analyzed (Participants) | 11 | 22
  Early Termination | 36.7 (0.18) | 36.6 (0.35)

25. Secondary Outcome: Vital Sign Examination: Blood Pressure (BP)
Description: Systolic BP: the measurement of the pressure when the heart is contracted (systole). The systolic pressure indicates the maximum amount of work/force the heart has to perform with each stroke in order to move blood through the arteries. Diastolic BP: the pressure in the large arteries during the relaxation of the left ventricle. The diastolic pressure indicates the amount of pressure the heart must overcome in order to generate the next beat.
Time Frame: Baseline (Day 1 0H), Week 2, 4, 6, 12, 16, Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here "overall number of participants analyzed" signifies participants who were evaluable for this measure; "number analyzed"=participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
millimeter of mercury (mmHg)
  Baseline Sitting Systolic BP | 125.4 (12.12) | 120.6 (12.23)
  Week 2 Sitting Systolic BP: number analyzed (Participants) | 27 | 27
  Week 2 Sitting Systolic BP | 121.9 (12.87) | 123.2 (14.05)
  Week 4 Sitting Systolic BP: number analyzed (Participants) | 27 | 26
  Week 4 Sitting Systolic BP | 121.4 (13.13) | 121.8 (15.56)
  Week 6 Sitting Systolic BP: number analyzed (Participants) | 23 | 25
  Week 6 Sitting Systolic BP | 117.9 (13.33) | 124.8 (14.38)
  Week 12 Sitting Systolic BP: number analyzed (Participants) | 13 | 7
  Week 12 Sitting Systolic BP | 120.4 (12.31) | 125.4 (11.39)
  Week 16 Sitting Systolic BP: number analyzed (Participants) | 12 | 6
  Week 16 Sitting Systolic BP | 124.0 (10.58) | 129.0 (17.38)
  Early Termination Sitting Systolic BP: number analyzed (Participants) | 11 | 22
  Early Termination Sitting Systolic BP | 114.5 (16.36) | 122.0 (17.12)
  Baseline Sitting Diastolic BP | 73.7 (8.71) | 75.0 (7.49)
  Week 2 Sitting Diastolic BP: number analyzed (Participants) | 27 | 27
  Week 2 Sitting Diastolic BP | 73.9 (8.07) | 75.6 (11.90)
  Week 4 Sitting Diastolic BP: number analyzed (Participants) | 27 | 26
  Week 4 Sitting Diastolic BP | 74.1 (9.48) | 73.2 (8.91)
  Week 6 Sitting Diastolic BP: number analyzed (Participants) | 23 | 25
  Week 6 Sitting Diastolic BP | 71.7 (9.55) | 75.3 (9.63)
  Week 12 Sitting Diastolic BP: number analyzed (Participants) | 13 | 7
  Week 12 Sitting Diastolic BP | 74.2 (8.07) | 78.4 (3.51)
  Week 16 Sitting Diastolic BP: number analyzed (Participants) | 12 | 6
  Week 16 Sitting Diastolic BP | 78.8 (9.09) | 80.2 (7.22)
  Early Termination Sitting Diastolic BP: number analyzed (Participants) | 11 | 22
  Early Termination Sitting Diastolic BP | 72.2 (13.26) | 72.9 (9.93)

26. Secondary Outcome: Vital Sign Examination: Respiratory Rate
Description: Respiration rate measured as number of breaths taken per minute.
Time Frame: Baseline (Day 1, 0H), Week 2, 4, 6, 12, 16, Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here "overall number of participants analyzed" signifies participants who were evaluable for this measure. "Number analyzed"=participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
breaths per minute
  Baseline | 15.5 (2.92) | 16.9 (2.61)
  Week 2: number analyzed (Participants) | 27 | 27
  Week 2 | 16.0 (3.52) | 16.8 (3.01)
  Week 4: number analyzed (Participants) | 27 | 27
  Week 4 | 15.6 (3.46) | 16.0 (3.04)
  Week 6: number analyzed (Participants) | 23 | 25
  Week 6 | 15.9 (3.28) | 16.1 (2.96)
  Week 12: number analyzed (Participants) | 13 | 7
  Week 12 | 14.7 (3.71) | 14.4 (2.99)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 15.1 (2.64) | 14.0 (2.45)
  Early Termination: number analyzed (Participants) | 11 | 22
  Early Termination | 16.4 (3.29) | 16.7 (2.78)

27. Secondary Outcome: Vital Sign Examination: Heart Rate
Description: Heart rate is the number of heart beats per minute.
Time Frame: Baseline (Day 1, 0H), Week 2, 4, 6, 12, 16, and Early Termination (up to 113 days)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
beats per minute
  Baseline | 82.1 (12.10) | 82.6 (12.85)
  Week 2: number analyzed (Participants) | 27 | 27
  Week 2 | 80.4 (13.10) | 81.3 (14.11)
  Week 4: number analyzed (Participants) | 27 | 27
  Week 4 | 78.5 (10.56) | 79.7 (12.23)
  Week 6: number analyzed (Participants) | 23 | 25
  Week 6 | 77.4 (10.01) | 80.1 (15.22)
  Week 12: number analyzed (Participants) | 13 | 7
  Week 12 | 78.2 (11.02) | 72.9 (10.04)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 85.3 (8.87) | 75.8 (12.94)
  Early Termination: number analyzed (Participants) | 11 | 22
  Early Termination | 79.2 (8.57) | 82.9 (17.26)

28. Secondary Outcome: Body Weight of Participants
Time Frame: Baseline, Week 6, 16 and Early Termination (up to 113 days)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 30
Kilogram (Kg)
  Baseline | 68.5 (11.98) | 72.6 (17.35)
  Week 6: number analyzed (Participants) | 23 | 24
  Week 6 | 67.4 (13.03) | 74.3 (17.67)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 66.5 (10.91) | 76.0 (14.60)
  Early Termination | 64.6 (12.12) | 73.1 (18.02)

29. Secondary Outcome: Number of Participants With Abnormal Laboratory Examination
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit (<0.8*lower limit of normal [LLN]); red blood cell count (<0.8*LLN); platelets (<0.5*LLN or >1.75* upper limit of normal [ULN]); leucocytes (<0.6*LLN or >1.5*ULN); lymphocytes, total neutrophils (<0.8*LLN or >1.2*ULN); basophils, eosinophils, monocytes (>1.2*ULN); total bilirubin (>1.5* ULN); aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase (>3*ULN); creatinine, blood urea nitrogen (>1.3*ULN); glucose (<0.6*LLN or >1.5*ULN); uric acid (>1.2*ULN); sodium (<0.95*LLN or 1.05*ULN); potassium, calcium, chloride, bicarbonate (<0.9*LLN or 1.1*ULN); albumin, total protein (<0.8*LLN or 1.2*ULN); urine analysis. Total number of participants without regards to baseline abnormality was summarized.
Time Frame: Baseline up to Week 16, Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here "overall number of participants analyzed" signifies those participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 27 | 29
Participants | 27 | 29

30. Secondary Outcome: Number of Participants With Anti-drug Antibodies
Description: Human serum samples were analyzed using electrochemiluminescent (ECL) immunoassay for the presence of anti-tanezumab antibodies. Same participant may have positive (titer value >=4.32) anti-tanezumab antibodies result at more than 1 time point.
Time Frame: Baseline (Day 1), Week 4, 6, 12, 16
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure. 'number analyzed'=participants evaluable at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab
Number analyzed (Participants) | 29
Participants
  Baseline: number analyzed (Participants) | 27
  Baseline | 0
  Week 4: number analyzed (Participants) | 26
  Week 4 | 1
  Week 6: number analyzed (Participants) | 22
  Week 6 | 0
  Week 12: number analyzed (Participants) | 11
  Week 12 | 0
  Week 16: number analyzed (Participants) | 23
  Week 16 | 1

31. Secondary Outcome: Electrocardiogram Examination
Description: ECG intervals included: RR (the time interval between consecutive heart beats), PR (time between the onset of atrial depolarization and the onset of ventricular depolarization), QRS (represented ventricular depolarization) and QT (time corresponding to the beginning of depolarization to repolarization of the ventricles), QTcF (QT interval corrected using Fridericia's formula [FF]), QTcB interval (QT interval corrected using Bazett's formula [BF]).
Time Frame: Baseline (Pre-dose and 1 hour Post-dose), Week 4, 16, Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here "overall number of participants analyzed" signifies participants who were evaluable for this measure; "number analyzed" =participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 28 | 30
millisecond (msec)
  Baseline Pre-dose RR interval | 742.7 (146.23) | 767.7 (153.09)
  Baseline 1 hour Post-dose RR interval: number analyzed (Participants) | 27 | 25
  Baseline 1 hour Post-dose RR interval | 774.9 (143.62) | 792.5 (157.81)
  Week 4 RR interval: number analyzed (Participants) | 26 | 25
  Week 4 RR interval | 774.1 (161.87) | 777.2 (161.81)
  Week 16 RR interval: number analyzed (Participants) | 12 | 6
  Week 16 RR interval | 805.4 (143.66) | 828.8 (150.78)
  Early Termination RR interval: number analyzed (Participants) | 10 | 22
  Early Termination RR interval | 805.0 (164.26) | 760.2 (152.61)
  Baseline Pre-dose PR interval: number analyzed (Participants) | 26 | 30
  Baseline Pre-dose PR interval | 162.2 (27.83) | 151.6 (15.82)
  Baseline 1 hour Post-dose PR interval: number analyzed (Participants) | 25 | 25
  Baseline 1 hour Post-dose PR interval | 163.6 (22.66) | 153.1 (18.26)
  Week 4 PR interval: number analyzed (Participants) | 24 | 25
  Week 4 PR interval | 162.2 (27.29) | 150.0 (17.44)
  Week 16 PR interval: number analyzed (Participants) | 24 | 25
  Week 16 PR interval | 169.7 (32.67) | 145.4 (16.27)
  Early Termination PR interval: number analyzed (Participants) | 9 | 22
  Early Termination PR interval | 164.0 (20.99) | 151.6 (17.60)
  Baseline Pre-dose QRS complex | 89.5 (10.53) | 93.7 (10.60)
  Baseline 1 hour Post-dose QRS complex: number analyzed (Participants) | 26 | 25
  Baseline 1 hour Post-dose QRS complex | 90.6 (10.54) | 94.0 (11.53)
  Week 4 QRS complex: number analyzed (Participants) | 26 | 25
  Week 4 QRS complex | 89.0 (9.97) | 92.2 (10.28)
  Week 16 QRS complex: number analyzed (Participants) | 12 | 6
  Week 16 QRS complex | 87.6 (11.93) | 94.5 (9.12)
  Early Termination QRS complex: number analyzed (Participants) | 10 | 22
  Early Termination QRS complex | 88.7 (10.33) | 93.0 (11.10)
  Baseline Pre-dose QT interval: number analyzed (Participants) | 27 | 30
  Baseline Pre-dose QT interval | 375.6 (33.19) | 384.6 (38.26)
  Baseline 1 hour Post-dose QT interval: number analyzed (Participants) | 24 | 25
  Baseline 1 hour Post-dose QT interval | 388.9 (34.08) | 389.9 (36.38)
  Week 4 QT interval: number analyzed (Participants) | 26 | 25
  Week 4 QT interval | 383.7 (36.19) | 384.6 (38.33)
  Week 16 QT interval: number analyzed (Participants) | 11 | 6
  Week 16 QT interval | 386.2 (25.93) | 394.2 (33.98)
  Early Termination QT interval: number analyzed (Participants) | 10 | 22
  Early Termination QT interval | 392.3 (42.72) | 385.8 (34.97)
  Baseline Pre-dose QTCB interval BF: number analyzed (Participants) | 27 | 30
  Baseline Pre-dose QTCB interval BF | 437.9 (22.08) | 441.6 (23.19)
  Baseline 1hour Post-dose QTCB interval BF: number analyzed (Participants) | 24 | 25
  Baseline 1hour Post-dose QTCB interval BF | 438.4 (19.46) | 440.7 (23.10)
  Week 4 QTCB interval BF: number analyzed (Participants) | 26 | 25
  Week 4 QTCB interval BF | 439.5 (24.83) | 439.0 (22.47)
  Week 16 QTCB interval BF: number analyzed (Participants) | 11 | 6
  Week 16 QTCB interval BF | 435.1 (22.31) | 434.9 (13.33)
  Early Termination QTCB interval BF: number analyzed (Participants) | 10 | 22
  Early Termination QTCB interval BF | 440.5 (24.86) | 445.5 (23.89)
  Baseline Pre-dose QTCB interval FF: number analyzed (Participants) | 27 | 30
  Baseline Pre-dose QTCB interval FF | 415.6 (19.50) | 421.3 (22.97)
  Baseline 1hour Post-dose QTCB interval FF: number analyzed (Participants) | 24 | 25
  Baseline 1hour Post-dose QTCB interval FF | 420.8 (20.05) | 422.7 (21.73)
  Week 4 QTCB interval FF: number analyzed (Participants) | 26 | 25
  Week 4 QTCB interval FF | 419.5 (21.64) | 419.6 (22.07)
  Week 16 QTCB interval FF: number analyzed (Participants) | 11 | 6
  Week 16 QTCB interval FF | 417.7 (15.59) | 420.6 (14.71)
  Early Termination QTCB interval FF: number analyzed (Participants) | 10 | 22
  Early Termination QTCB interval FF | 423.3 (25.07) | 424.1 (20.93)

32. Secondary Outcome: Electrocardiogram Examination: Heart Rate
Description: Standard 12-lead ECG performed after participant had rested quietly for at least 10 minutes in a supine position was measured. The time interval between consecutive heart beats [RR interval] (in beats per minute [bpm]) was used to calculate heart rate.
Time Frame: Baseline (Pre-dose and 1 hour Post-dose), Week 4, 16, Early Termination (up to 113 days)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo). Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure; "number analyzed"=participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 28 | 30
bpm
  Baseline Pre-dose | 84.0 (16.89) | 81.1 (15.33)
  Baseline 1 hour Post-dose: number analyzed (Participants) | 27 | 25
  Baseline 1 hour Post-dose | 80.1 (15.33) | 78.5 (14.57)
  Week 4: number analyzed (Participants) | 26 | 25
  Week 4 | 80.9 (16.75) | 80.2 (14.99)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 77.0 (13.69) | 74.4 (12.71)
  Early Termination: number analyzed (Participants) | 10 | 22
  Early Termination | 77.6 (16.25) | 81.9 (15.64)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tanezumab | Placebo
Serious Adverse Events (participants affected / at risk) | 7/29 | 4/30
Other Adverse Events (participants affected / at risk) | 14/29 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=29) | Placebo (N=30)
Cardiac failure acute (Cardiac disorders) | 1 | 0
Proctitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=29) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Somnolence (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.